CLINICAL TRIAL: NCT03205852
Title: Do we Really Allow Patient Decision-making in Rotator Cuff Surgery? A Prospective Randomized Study
Brief Title: Patients Decision-making in Rotator Cuff Surgery
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Chief Clinic Upper Limb, Hospital del Mar
Other Study IDs: 2014/5625/I
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Rotator Cuff Disease
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A (benefit-inform): filling questionnaire based on benefits of surgery
  Interventions: Other: questionnaire
- group B (side effect-inform): filling questionnaire based on side-effects of surgery
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — fulfillment of questionnaire

SUMMARY:
The objective of this study was to evaluate the effect on patient treatment decision-making if information was given based on the benefit or on the side effect in rotator cuff disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with rotator cuff tears at their first clinical visit

Exclusion Criteria:

* patients with a previous shoulder surgery, patients with worker's compensation and patients who were unwilling to participate and thereby not sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosis of rotator cuff tears documented by MRI
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2014-09-05 (Actual); Study Completion 2014-12-29 (Actual)

PRIMARY OUTCOMES:
questionnaire of surgery decision | immediate
  two proposals for surgery based on information given to the patient

SECONDARY OUTCOMES:
Constant Score | immediate
  functional evaluation of shoulder function

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Torrens C, Miquel J, Santana F. Do we really allow patient decision-making in rotator cuff surgery? A prospective randomized study. J Orthop Surg Res. 2019 Apr 29;14(1):116. doi: 10.1186/s13018-019-1157-2. PMID 31036041